CLINICAL TRIAL: NCT02978482
Title: A Phase 1/2 Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of Durvalumab (MEDI4736) in Combination With Tremelimumab in Chinese Patients With Advanced Malignancies
Brief Title: A Phase 1/2 Study of Durvalumab(MEDI4736) and Tremelimumab in Chinese Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419AC00006
Record Dates: First submitted 2016-11-08; First posted 2016-12-01 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Advanced Malignancy
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- durvalumab (Experimental): durvalumab alone
  Interventions: Drug: durvalumab
- durvalumab+tremelimumab (Experimental): durvalumab plus tremelimumab
  Interventions: Drug: tremelimumab + durvalumab

INTERVENTIONS:
Drug: durvalumab — durvalumab (MEDI4736) 20mg/kg via IV infusion every 4 weeks until confirmed disease progression or unacceptable toxicity
  Arms: durvalumab
Drug: tremelimumab + durvalumab — 20 mg/kg durvalumab (MEDI4736) via IV infusion q4w and 1 mg/kg tremelimumab via IV infusion q4w for up to 4 doses/cycles, and then continue 20 mg/kg durvalumab (MEDI4736) q4w starting on Week 16 for up to confirmed disease progression
  Arms: durvalumab+tremelimumab

SUMMARY:
A Phase 1/2 Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of Durvalumab (MEDI4736) in combination with tremelimumab in Chinese Patients with Advanced Malignancies

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Male or female, aged at least 18 years
* For Phase 1 PK cohort:

Patients with histologically or cytologically confirmed advanced and/or metastatic solid tumors other than HCC refractory or intolerable to existing standard of treatment

For Phase 2 cohort:

For nasopharyngeal carcinoma:

Patients with histologically or cytologically confirmed nasopharyngeal carcinoma must have locally advanced or metastatic disease progressed on or after at least 1 chemotherapy regimen with or without radiotherapy.

* ONLY FOR PHASE 2 PORTION: mandatory tumor sample
* No prior exposure to immune-mediated therapy including, but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
* Life expectancy ≥12 weeks at Day 1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* At least 1 lesion that can be accurately measured at baseline, and that is suitable for repeated measurements as per RECIST 1.1 guidelines.
* Adequate organ and marrow function
* Hemoglobin ≥9 g/dL Absolute neutrophil count ≥1.0 × 109 /L Platelet count ≥75 × 109/L Total serum bilirubin ≤1.5×upper limit of normal (ULN) ALT and AST ≤2.5×ULN; for patients with hepatic metastases, ALT and AST ≤5×ULN Calculated creatinine clearance >40 mL/min as determined by Cockcroft-Gault (using actual body weight), or by measured 24-hour urine collection for determination of creatinine clearance.
* Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients.
* Exclusion Criteria:
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable. Note: Local treatment of isolated lesions for palliative intent is acceptable (eg, local surgery or radiotherapy).
* Receipt of last dose of an approved (marketed) anticancer therapy (chemotherapy, targeted therapy, biologic therapy, mAbs, etc) within 21 days prior to the first dose of study treatment. If sufficient washout time has not occurred due to the schedule or PK properties of an agent, a longer washout period will be required, as agreed upon by AstraZeneca and the Investigator.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation
* Any unresolved toxicity National Cancer Institute (NCI) CTCAE Version 4.03 Grade ≥2 from previous anticancer therapy
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc).
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of another primary malignancy
* History of leptomeningeal carcinomatosis
* Brain metastases or spinal cord compression unless asymptomatic or treated and stable off steroids and anti-convulsants for at least 14 days prior to study treatment.
* QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated.
* History of active primary immunodeficiency
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus .
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab (MEDI4736) or tremelimumab.
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of IP.
* Female patients who are pregnant or breast-feeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab (MEDI4736) plus tremelimumab combination therapy or 90 days after the last dose of durvalumab (MEDI4736) monotherapy.
* Known allergy or hypersensitivity to IP or any IP excipient, or to other humanized mAbs
* Prior randomisation or treatment in a previous durvalumab (MEDI4736) and/or tremelimumab clinical study regardless of treatment arm assignment
* NSCLC patients have history of interstitial lung disease

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | approximately 6 months after the last evaluable patient in Phase 1 portion is first dosed
  Only for phase 1 portion of the study
Trough plasma concentration (Ctrough) | approximately 6 months after the last evaluable patient is first dosed in phase 1 portion
  Only for phase 1 portion of the study
Area under the plasma drug concentration-time curve from time zero to Day 28 post-dose (AUC 0-28) | approximately 6 months after the last evaluable patient is first dosed in phase 1 portion
  Only for phase 1 portion of the study
Adverse event | Approximately 12 months after the last evaluable patient from Ph 1 is 1st dosed or the last patient has withdrawn from study or the study discontinued by Sponsor
Objective response rate (ORR) | Approximately 12 months after the last evaluable patient is dosed, or the last patient has withdrawn from the study or the study is discontinued by the sponsor.
  Only for phase 2 portion of the study (Phase 2 part withdrawn without initiation)

SECONDARY OUTCOMES:
Anti-drug antibody (ADA) | approximately 12 months after the last evaluable patient is first dosed, or the last patient has withdrawn from the study, or the study is discontinued by the Sponsor
Anti-drug antibody neutralizing antibodies (ADA nAB) | approximately 12 months after the last evaluable patient is first dosed, or the last patient has withdrawn from the study, or the study is discontinued by the Sponsor
Complete response/Partial response/Stable disease/Progressive disease | approximately 6 months after the last evaluable patient is first dosed in phase 1 portion
  Only for phase 1 portion of the study
Overall survival (OS) | approximately 12 months after the last evaluable patient is first dosed, or the last patient has withdrawn from the study, or the study is discontinued by the Sponsor
  Only for phase 2 portion of the study (Phase 2 part withdrawn without initiation)

OTHER OUTCOMES:
PD-L1 status | through study completion, an average of 2 years
  Only for phase 2 portion of the study (Phase 2 part withdrawn without initiation)
CD8+ T cells | through study completion, an average of 2 years
  Only for phase 2 portion of the study (Phase 2 part withdrawn without initiation)
IFNγ | through study completion, an average of 2 years
  Only for phase 2 portion of the study (Phase 2 part withdrawn without initiation)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute; Urban Scheuring, Study Director — AstraZeneca GMD IO, Melbourn Science Park, Melbourn, Royston, Hertfordshire, SG8 6HB, UK
Locations (1):
- Research Site, Changchun, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search